CLINICAL TRIAL: NCT02888730
Title: Efficacy of Antibiotic (Tobramycin) Delivered by Nebulized Sonic Aerosol for Chronic Rhinosinusitis Treatment of Cystic Fibrosis Patients: A Multicenter Double-blind Randomized Controlled Trial
Brief Title: Tobramycin Delivered by Nebulized Sonic Aerosol for Chronic Rhinosinusitis Treatment of Cystic Fibrosis Patients
Acronym: AVASMUC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No suffisant recruitment
Sponsor: Virginie ESCABASSE (Other)
Collaborators: Henri Mondor University Hospital (Other)
Responsible Party: Sponsor-Investigator, Virginie ESCABASSE, MD, PhD, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVASMUC
Record Dates: First submitted 2016-06-22; First posted 2016-09-05 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis; Rhinosinusitis; Lung Diseases
Keywords: cystic fibrosis; chronic rhinosinusitis; Lung Diseases; tobramycin; nebulized sonic aerosol therapy
MeSH Terms: conditions — Cystic Fibrosis; Rhinosinusitis; Lung Diseases | interventions — Tobramycin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobramycin nebulized nasally (Experimental): Nebulized Tobramycin, one bulb (tobramycin 300 mg and sodium chloride 11.25 mg) nasally twice a day for 15 days
  Interventions: Drug: Tobramycin nebulized nasally
- Physiologic serum nebulized nasally (Placebo Comparator): Nebulized sodium chloride 0.9%, one bulb twice a day nasally for 15 days
  Interventions: Drug: Physiologic serum nebulized nasally

INTERVENTIONS:
Drug: Tobramycin nebulized nasally — Two sonic nebulizations per day will be realized by patients: morning and evening during 15 days. There should be a maximum of 12 hours between the 2 doses but shall not be less than 6 hours. The dosage should not be adjusted to body weight. All patients will receive one ampoule of tobramycin twice a dayAmpoules of tobramycin are filled by 5 ml containing 300 mg of tobramycin and 11.25 mg of sodium chloride. Bulb should be employed in nebulizer and administered by the inhalation route approximately 15 minutes to complete.Antibiotic retained for the study, tobramycin is manufactured by the "Pharmacie à Usage Interne" of the Henri Mondor Hospital. The study's product will be prepared with Base Tobramycin and excipients in accordance with TOBI's composition.
  Other Names: Tobramycin
  Arms: Tobramycin nebulized nasally
Drug: Physiologic serum nebulized nasally — Two sonic nebulizations per day will be realized by patients: morning and evening during 15 days. There should be a maximum of 12 hours between the 2 doses but shall not be less than 6 hours. The dosage should not be adjusted to body weight. All patients will receive one ampoule of placebo (Nacl 0.9%) twice a day.Ampoules of placebo are filled by 5 ml containing of sodium chloride. Bulb should be employed in nebulizer and administered by the inhalation route approximately 15 minutes to complete. Placebo for the study is manufactured by the "Pharmacie à Usage Interne" of the Henri Mondor Hospital. Patients in placebo arm will receive 5ml of sodium chloride with the same color (light yellow transparent) as tobramycin
  Other Names: sodium chloride 0.9%
  Arms: Physiologic serum nebulized nasally

SUMMARY:
Patients with cystic fibrosis frequently develop chronic rhinosinusitis. Bacterial colonization is facilitated by a reduced mucociliary function and some previous studies suggest that the microbiology of the upper airways might influence the microbiology of the lower airway. The aim of this randomized control study is to demonstrate efficacy of antibiotic delivered by nebulized sonic aerosol therapy to decrease the bacterial load in sinuses and medium ostia and to improve the sino-nasal symptoms and endoscopic scores, quality of life and lung function

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common lethal autosomal recessive disorder in the Caucasian population affecting ~1:3000 children, with a carrier frequency of 1:25. It is a multisystem disorder where pulmonary and sinonasal involvements occur in 90-100% of patients, and up to 86% of children have nasal polyps . Patients with CF develop chronic rhinosinusitis (CRS) due to the defect in the cystic fibrosis Transmembrane Regulator (CFTR) protein. The membrane lining the paranasal sinuses and the nose is identical to the membrane lining the lungs. As in lower airways (LAW) the defect CFTR protein result in viscous mucus . Consequently mucociliary function is reduced, which facilitates bacterial colonization and eventually infection leading to rhinosinusitis . In the past decades infection of the lower airways was the most prominent focus in treatment protocols for CF. Over the years infection of the upper airways (UAW) gradually gained more attention in CF.

Previous research in the microbiology of the upper airways (UAW) in CF displayed that Haemophilus influenzae, Pseudomonas aeruginosa and Staphylococcus aureus were most frequently cultures from the UAW . Since several studies showed concordance between organisms in the UAW and the LAW in CF, the hypothesis evolved that the UAW might influence the patient pulmonary status . Moreover, comparison of UAW and and LAW cultures in CF adult patients showed that Pseudomonas aeruginosa can be cultured from the UAW after eradication therapy which may suggest persistence of Pseudomonas aeruginosa in the UAW . This problem is highlighted in double lung transplant where UAW also appears as a protective niche of adapted clones of bacteria, which can intermittently spread this pathogen to the lung.

CRS treatment in CF patients is based on daily nasal lavages but above all on local or systemic antibiotic treatments to eradicate bacteria in sinuses . Local therapy is favoured in CRS treatment of CF patients to avoid antibiotic side effects, changing organisms or resistance patterns. Sonic aerosol therapy with antibiotics for 15 days is commonly used for CRS in non CF patients to improve sinonasal symptoms and reduce purulent secretions as sound addition in pneumatic aerosol in head corpse's models creates an acoustic pressure at the ostia to improve the aerosol penetration in maxillary sinuses . However its efficacy on bacterial carrying in sinuses is not proved . At the opposite, efficacy of aerosol of tobramycin to LAW was proved in CF patients with a decrease of the density of Pseudomonas aeruginosa, an improvement of FEV, and fewer pulmonary exacerbations .

At the present time, efficacy of antibiotic (tobramycin) delivered by nebulized sonic aerosol for CRS treatment of CF patients is unknown particularly on bacterial carrying.

The aim of this study is to demonstrate that nebulized sonic aerosol therapy with tobramycin in Cystic Fibrosis patients decreases significantly bacterial carrying in sinuses, sinus ostia of middle meatus and sputum compared to nebulized sonic aerosol therapy with placebo and that nebulized sonic aerosol therapy improves sino-nasal symptoms and endoscopic scores, quality of life and lung function.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 7 years followed in the 6 CRCM centers (Créteil, Marseille, Nantes, Toulouse, Clermont-Ferrand and Nice). We choose to enroll children aged 7 years or more because as they have a better adherence to nebulization treatment than younger children.
* Diagnosis of cystic fibrosis confirmed by sweat test (>60mmol/L) and/or the identification of two CF-causing mutations
* Confirmed chronic rhinosinusitis by Ear Nose and Throat doctor by endoscopic examination: bilateral mucopurulent secretions at middle meatus present longer than 12 weeks with or without nasal polyps
* Positive bacteria susceptibility to tobramycin in samples from middle meatus
* Susceptibility of bacteria to tobramycin confirmed
* Pulmonary examination before enrollment
* Written informed consent obtained at enrollment for all patients (consent of minor's parent for children)
* Social security affiliation

Exclusion Criteria:

* - Oral antibiotic therapy one month before enrollment
* enrollment in another protocol with antibiotic
* Ongoing aerosolized tobramycin for endobronchial infection to avoid an overlap between treatment for lung and treatment for sinusitis
* Abnormal auditory acuity (decrease of 20dB in auditory acuity)
* Hypersensibility or allergenecity of aminoglycosides
* FEV < 25% or FVC of 40% or more of the value predicted for height
* Transplant patient or patient on transplant list
* Patient under nasal oxygen or under noninvasive ventilation
* Pregnant woman
* Breast-feeding
* No Social security affiliation
* Informed consent non obtained at enrollment for all patients (consent of minor's parent for children)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Density of bacteria (in CFU/g log10) in sinus ostia of middle meatus samples at day 15 | 15 days

SECONDARY OUTCOMES:
density of bacteria (in CFU/g log10) in sinus ostia of middle meatus samples at day 30 and 90 | day 30 and day 90
Minimum inhibitor concentration of sputum bacteria to antibiotics | day 15, 30 and 90
Minimum inhibitor concentration of sputum bacteria to tobramycin | day 90
Force Vital capacity (FCV) in both groups | day 0 and day 30
Forced Expiratory Volume in one second (FEV1) in both groups | day 0 and day 30
nasal obstruction at day 90 compared to baseline | day 0, 15, 30 and 90
rhinorrhea compared to baseline | day 0, 15, 30 and 90
mucopurulent secretions compared to baseline | day 0, 15, 30 and 90
facial pain compared to baseline | day 0, 15, 30 and 90
dysosmia compared to baseline | day 0, 15, 30 and 90
Nasal endoscopic scores compared to baseline in both groups | day 0, 15, 30 and 90
Score of the SM5 quality of life questionnaire in both groups | day 0, 15, 30 and 90
Score of the SNOT20 quality of life questionnaire in both groups | day 0, 15, 30 and 90
Hearing perception of the intensity (in db) and tone (Hz) of sound waves | day 0 and day 30

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Escabasse, MD, Principal Investigator — Creteil Hospital center (CHIC)
Locations (6):
- France (6):
  - Centre Hospitalier Universitaire de Clermont ferrand, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Universitaire de la Timone, Marseille
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Centre Hosiptalier de Nice, Nice
  - Centre Hospitalier Universitaire de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aanaes K, von Buchwald C, Hjuler T, Skov M, Alanin M, Johansen HK. The effect of sinus surgery with intensive follow-up on pathogenic sinus bacteria in patients with cystic fibrosis. Am J Rhinol Allergy. 2013 Jan;27(1):e1-4. doi: 10.2500/ajra.2013.27.3829. PMID 23406585
- [Background] Berkhout MC, Rijntjes E, El Bouazzaoui LH, Fokkens WJ, Brimicombe RW, Heijerman HG. Importance of bacteriology in upper airways of patients with Cystic Fibrosis. J Cyst Fibros. 2013 Sep;12(5):525-9. doi: 10.1016/j.jcf.2013.01.002. Epub 2013 Jan 26. PMID 23357546
- [Background] Boucher RC. Human airway ion transport. Part one. Am J Respir Crit Care Med. 1994 Jul;150(1):271-81. doi: 10.1164/ajrccm.150.1.8025763. No abstract available.
- [Background] Boucher RC. Human airway ion transport. Part two. Am J Respir Crit Care Med. 1994 Aug;150(2):581-93. doi: 10.1164/ajrccm.150.2.8049852. No abstract available.
- [Background] Coste A, Gilain L, Roger G, Sebbagh G, Lenoir G, Manach Y, Peynegre R. Endoscopic and CT-scan evaluation of rhinosinusitis in cystic fibrosis. Rhinology. 1995 Sep;33(3):152-6. PMID 8560168
- [Background] Digoy GP, Dunn JD, Stoner JA, Christie A, Jones DT. Bacteriology of the paranasal sinuses in pediatric cystic fibrosis patients. Int J Pediatr Otorhinolaryngol. 2012 Jul;76(7):934-8. doi: 10.1016/j.ijporl.2012.02.043. Epub 2012 Apr 17. PMID 22513080
- [Background] Durand M, Pourchez J, Aubert G, Le Guellec S, Navarro L, Forest V, Rusch P, Cottier M. Impact of acoustic airflow nebulization on intrasinus drug deposition of a human plastinated nasal cast: new insights into the mechanisms involved. Int J Pharm. 2011 Dec 12;421(1):63-71. doi: 10.1016/j.ijpharm.2011.09.023. Epub 2011 Sep 21. PMID 21963472
- [Background] Durand M, Le Guellec S, Pourchez J, Dubois F, Aubert G, Chantrel G, Vecellio L, Hupin C, De Gersem R, Reychler G, Pitance L, Diot P, Jamar F. Sonic aerosol therapy to target maxillary sinuses. Eur Ann Otorhinolaryngol Head Neck Dis. 2012 Oct;129(5):244-50. doi: 10.1016/j.anorl.2011.09.002. Epub 2012 Aug 24. PMID 22921302
- [Background] Gysin C, Alothman GA, Papsin BC. Sinonasal disease in cystic fibrosis: clinical characteristics, diagnosis, and management. Pediatr Pulmonol. 2000 Dec;30(6):481-9. doi: 10.1002/1099-0496(200012)30:63.0.co;2-n. PMID 11109061
- [Background] Hansen SK, Rau MH, Johansen HK, Ciofu O, Jelsbak L, Yang L, Folkesson A, Jarmer HO, Aanaes K, von Buchwald C, Hoiby N, Molin S. Evolution and diversification of Pseudomonas aeruginosa in the paranasal sinuses of cystic fibrosis children have implications for chronic lung infection. ISME J. 2012 Jan;6(1):31-45. doi: 10.1038/ismej.2011.83. Epub 2011 Jun 30. PMID 21716309
- [Background] Kahl BC, Duebbers A, Lubritz G, Haeberle J, Koch HG, Ritzerfeld B, Reilly M, Harms E, Proctor RA, Herrmann M, Peters G. Population dynamics of persistent Staphylococcus aureus isolated from the airways of cystic fibrosis patients during a 6-year prospective study. J Clin Microbiol. 2003 Sep;41(9):4424-7. doi: 10.1128/JCM.41.9.4424-4427.2003. PMID 12958283
- [Background] Knowles MR, Robinson JM, Wood RE, Pue CA, Mentz WM, Wager GC, Gatzy JT, Boucher RC. Ion composition of airway surface liquid of patients with cystic fibrosis as compared with normal and disease-control subjects. J Clin Invest. 1997 Nov 15;100(10):2588-95. doi: 10.1172/JCI119802. PMID 9366574
- [Background] Konstan MW, Morgan WJ, Butler SM, Pasta DJ, Craib ML, Silva SJ, Stokes DC, Wohl ME, Wagener JS, Regelmann WE, Johnson CA; Scientific Advisory Group and the Investigators and Coordinators of the Epidemiologic Study of Cystic Fibrosis. Risk factors for rate of decline in forced expiratory volume in one second in children and adolescents with cystic fibrosis. J Pediatr. 2007 Aug;151(2):134-9, 139.e1. doi: 10.1016/j.jpeds.2007.03.006. Epub 2007 Jun 22. PMID 17643762
- [Background] Mainz JG, Naehrlich L, Schien M, Kading M, Schiller I, Mayr S, Schneider G, Wiedemann B, Wiehlmann L, Cramer N, Pfister W, Kahl BC, Beck JF, Tummler B. Concordant genotype of upper and lower airways P aeruginosa and S aureus isolates in cystic fibrosis. Thorax. 2009 Jun;64(6):535-40. doi: 10.1136/thx.2008.104711. Epub 2009 Mar 11. PMID 19282318
- [Background] Ramsey BW, Dorkin HL, Eisenberg JD, Gibson RL, Harwood IR, Kravitz RM, Schidlow DV, Wilmott RW, Astley SJ, McBurnie MA, et al. Efficacy of aerosolized tobramycin in patients with cystic fibrosis. N Engl J Med. 1993 Jun 17;328(24):1740-6. doi: 10.1056/NEJM199306173282403. PMID 8497284
- [Background] Regnis JA, Robinson M, Bailey DL, Cook P, Hooper P, Chan HK, Gonda I, Bautovich G, Bye PT. Mucociliary clearance in patients with cystic fibrosis and in normal subjects. Am J Respir Crit Care Med. 1994 Jul;150(1):66-71. doi: 10.1164/ajrccm.150.1.8025774.
- [Background] Robertson JM, Friedman EM, Rubin BK. Nasal and sinus disease in cystic fibrosis. Paediatr Respir Rev. 2008 Sep;9(3):213-9. doi: 10.1016/j.prrv.2008.04.003. Epub 2008 Jul 31. PMID 18694713
- [Background] Vaughan WC, Carvalho G. Use of nebulized antibiotics for acute infections in chronic sinusitis. Otolaryngol Head Neck Surg. 2002 Dec;127(6):558-68. doi: 10.1067/mhn.2002.129738. PMID 12501108
- [Background] Walter S, Gudowius P, Bosshammer J, Romling U, Weissbrodt H, Schurmann W, von der Hardt H, Tummler B. Epidemiology of chronic Pseudomonas aeruginosa infections in the airways of lung transplant recipients with cystic fibrosis. Thorax. 1997 Apr;52(4):318-21. doi: 10.1136/thx.52.4.318. PMID 9196512
- [Derived] Karanth TK, Karanth VKLK, Ward BK, Woodworth BA, Karanth L. Medical interventions for chronic rhinosinusitis in cystic fibrosis. Cochrane Database Syst Rev. 2022 Apr 7;4(4):CD012979. doi: 10.1002/14651858.CD012979.pub3. PMID 35390177